CLINICAL TRIAL: NCT07040072
Title: The Safety and Efficacy of Finotonlimab Combined With Stapokibart in the Treatment of Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma, a Phase Ib Study
Brief Title: Finotonlimab Combined With Stapokibart in the Treatment of Recurrent/Metastatic HNSCC
Acronym: LONG'E
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Keymed Biosciences Co.Ltd (Industry); Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR Sta-Fin (LONG'E)
Record Dates: First submitted 2025-04-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stapokibart and Finotonlimab (Experimental): Stapokibart, 600 mg for the first cycle, 300 mg for the second and third cycles, administered subcutaneously every three weeks, for a total of 3 doses.
  Finotonlimab 200 mg, administered intravenously once every three weeks, until disease progression or unacceptable toxicity.
  Interventions: Combination Product: Stapokibart and Finotonlimab

INTERVENTIONS:
Combination Product: Stapokibart and Finotonlimab — Receive the combination of Stapokibart and Finotonlimab in cycles 1-3, and maintain treatment with Finotonlimab in subsequent cycles.
  Stapokibart, 600mg for the first cycle, 300mg for the second and third cycles, administered subcutaneously every 3 weeks, for a total of 3 doses of Stapokibart; Finotonlimab 200mg, administered intravenously every 3 weeks until confirmed disease progression occurs according to the RECIST 1.1 imaging criteria (if the researcher determines that the subject can benefit from continuing PD-1 drug treatment, and the subject can tolerate the study treatment and agree, PD-1 drug can be continued and recorded in the study records), unacceptable toxic side effects, initiation of new anti-tumor treatment, withdrawal from the study or death (whichever occurs first), or reaching a maximum treatment period of 2 years.

SUMMARY:
This is a single-arm, phase Ib study involving HNSCC patients who had received first-line treatment with either PD-1 combined with platinum-based drugs or PD-1 monotherapy. The aim of the study is to evaluate the safety and efficacy of Finotonlimab in combination with Stapokibart in the treatment of recurrent/metastatic HNSCC patients.

DETAILED DESCRIPTION:
This study includes a total of 10 participants. Firstly, three participants will be enrolled to receive the combination therapy regimen. Safety observations will be conducted within 30 days after the third participant completes the third cycle of Stapokibart and Finotonlimab combination therapy. Based on the collected trial data, the investigators will evaluate and provide a safety report. If a major safety event or other factor affecting participant safety was identified, the treatment regimen will be re-evaluated before proceeding with further enrollment. Adjustments to administration frequency, dosage, and sample size can be made, or the trial can be terminated; If no safety concerns are identified, the remaining seven participants will be enrolled according to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the ICF;
2. Recurrent/metastatic HNSCC diagnosed histologically or cytologically in the oral, oropharyngeal, pharyngeal, and laryngeal regions;
3. Male/female, ≥ 18 years old, ECOG 0~1;
4. After PD-1 and platinum therapy, or PD-1 monotherapy, disease progression occurs within 12 weeks after the last ICI administration (as assessed by RECIST 1.1);
5. Target lesion (RECIST 1.1);
6. Previous PD-L1 expression test results may provide tissue for PD-L1 immunohistochemical testing;
7. Expected to survive for more than 3 months;
8. The main organ functions must meet the following requirements (laboratory test values within 7 days before enrollment must meet the following standards):

   * Blood routine examination: (No blood transfusion, no use of granulocyte colony-stimulating factor, no medication correction within 14 days before screening): a) Neutrophils ≥ 1.5 × 109/L; b) Platelets ≥ 75 × 109/L; c) Hemoglobin ≥ 90g/L; ② Biochemical examination: (No albumin transfusion within 14 days before screening): a) Blood creatinine ≤ 1.5 x upper limit of normal (ULN), or creatinine clearance rate>50 mL/min; b) Serum total bilirubin ≤ 1.5 × ULN; c) Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; ③ Coagulation function: a) International normalized ratio (INR) ≤ 2.3 or prothrombin time (PT) exceeding the normal control range ≤ 6 seconds.

Exclusion Criteria:

1. Suitable for local treatment;
2. Merge with other malignant tumors;
3. Brain metastasis;
4. If the toxicity does not recover to level 0-1 after surgery/radiotherapy/drug treatment, excluding chronic toxicity;
5. Allergic to known medication ingredients;
6. Major surgeries, radiation therapy (excluding palliative care), chemotherapy, immunotherapy, and biologics within 4 weeks prior to enrollment;
7. Received TKI, palliative surgery, and non-specific immunomodulatory therapy (such as thymosin and interferon) within 2 weeks before enrollment;
8. Received traditional Chinese patent medicines and simple preparations within one week before enrollment;
9. Use immunosuppressive drugs within 4 weeks before enrollment (excluding short-term, local, and physiological dose hormone therapy);
10. Patients with the following infection conditions:

    Active infections require systemic use of antibiotics; Active mycobacterium tuberculosis infection (i.e. tuberculosis infection); Hepatitis C virus antibody (HCV Ab) positive and hepatitis C virus ribonucleic acid (HCV-RNA) positive; Hepatitis B virus deoxyribonucleic acid (HBV-DNA) ≥ 1000 IU/mL; History of human immunodeficiency virus (HIV) infection or HIV antibody positivity during screening period.
11. Uncontrollable pleural effusion, abdominal effusion, and pericardial effusion;
12. Previous grade ≥ 3 irAE or grade ≥ 2 myocarditis;
13. Have a serious history of cardiovascular and cerebrovascular diseases, including but not limited to:

    Major cardiovascular and cerebrovascular diseases (such as congestive heart failure, acute myocardial infarction, unstable angina, stroke, transient ischemic attack, deep vein thrombosis or pulmonary embolism, etc.) occurred within 6 months before the first administration; Corrected QT interval (QTcF)>480 milliseconds; Echocardiography (ECHO) indicates that the subject's left ventricular ejection fraction (LVEF) is less than 50%; New York Heart Association (NYHA) heart function classification ≥ 2; Clinically uncontrollable hypertension (note: diastolic blood pressure ≥ 100mmHg or systolic blood pressure ≥ 160mmHg. If blood pressure is controlled with or without intervention, subjects can continue to be screened); Other cardiovascular and cerebrovascular diseases that have been evaluated by the researchers as unsuitable for participation in this study;
14. Active autoimmune diseases;
15. There is a significant risk of bleeding;
16. Receive a live vaccine within 4 weeks before enrollment;
17. During pregnancy or lactation, subjects with fertility do not receive contraceptive measures;
18. The presence of mental illness may affect the conduct of clinical trials;
19. History of organ transplantation or stem cell transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to 2 years
  Number of participants with AEs assessed by Common Terminology Criteria for Adverse Events v5.0.
Overall response rate (ORR) | Up to 2 years
  Percentage of participants with a confirmed best overall complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  The proportion of participants who achieve complete response (CR), partial response (PR), or stable disease (SD) as their best overall response, according to RECIST 1.1 criteria.
Progression free survival (PFS) | Up to 2 years
  PFS will be calculated from the first administration of Stapokibart to the date of documented disease progression, or death from any cause.
Duration of response (DOR) | Up to 2 years
  The time from the date of first response (CR or PR) to the date of progression of disease or death of any cause.

OTHER OUTCOMES:
Histopathological evaluation of tumor tissues | Up to 10 weeks
  Investigate changes in the proportions of Ki67-, p63-, and EGFR-positive cells in tumor specimens before and after treatment with Stapokibart and Finotonlimab.
Tumor-infiltrating immune cell subtypes | up to 10 weeks
  Evaluate changes in the proportions of T cells, B cells, natural killer cells, dendritic cells, macrophages and mast cells in tumor tissues before and after treatment.
Serum cytokine profiles | up to 10 weeks
  Assess changes in serum cytokine profiles before and after treatment, including IL-4, IL-13, IFN-γ, IL-17A, IL-8, IL-10, and other relevant cytokines.
Peripheral immune cell subtypes and activation status | up to 10 weeks
  Evaluate changes in the proportions and activation status of peripheral immune cell subtypes before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Study Chair — Beijing Tong-Ren hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China